CLINICAL TRIAL: NCT01216085
Title: An Exploratory Single Center Study of High-dose Treatment of Glivec® in Patients With Newly Diagnosed, Previously Untreated Chronic Myeloid Leukemia in Chronic Phase (CML-CP) Using Molecular Endpoints - TOPS (Tyrosine Kinase Inhibitor Optimization and Selectivity) Study
Brief Title: An Exploratory Study of High-dose Glivec in Patients With CML-CP Using Molecular Endpoints
Acronym: CML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571AKR23
Record Dates: First submitted 2010-09-27; First posted 2010-10-07 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2020-10

CONDITIONS: CML; Imatinib
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (1):
- imatinib (Experimental): Study patients will receive 400 mg twice daily oral administration in the morning and the evening.
  Interventions: Drug: high-dose imatinib

INTERVENTIONS:
Drug: high-dose imatinib — Study patients will receive 400 mg twice daily oral administration in the morning and the evening.

SUMMARY:
This study is locally amended study from CSTI571K2301 to evaluate the efficacy and safety of high-dose Glivec in Korean patients group with chronic phase of CML. Molecular response at 60 months after Glivec administration will be described.

ELIGIBILITY:
Inclusion Criteria:

1. TOPS(CSTI571K2301) participant patients who are taking Glivec more than 400 mg daily as 30 July, 2010, the close date of TOPS
2. Patients who provided written informed consent prior to participation to this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Major molecular response | 60 months
  Major molecular response achieved to Month 60 from the time of Glivec treatment

SECONDARY OUTCOMES:
progression-free survival | until 60 months
  Besides Complete molecular response, complete and major cytogenetic response achieved, event-free survival, and survival without progression to AP/BC achieved to Month 60 from the time of Glivec treatment, Progression-free survival will be evaluated.
number of adverse events | until 60 months
  compliance status and adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Wook Kim, MD, PhD, Principal Investigator — Catholic Medical Center
Locations (1):
- Novartis Investigational Site, Seoul, South Korea